CLINICAL TRIAL: NCT04486027
Title: Can Cytokines be Used as an Activation Marker in Rheumatoid Arthritis
Brief Title: Can Cytokines be Used as an Activation Marker
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Selim Nalbant, Prof, Maltepe University
Other Study IDs: 2017/900/19
Record Dates: First submitted 2020-07-13; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: c reactive protein; Erythrocyte sedimentation rate; DAS-28; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: Healthy individuals not smoking, not using Disease-Modifying Anti-Rheumatic Drugs (DMARD) and/or anti-inflammatory drugs other than cortisol and methotrexate, not receiving chemotherapy, not being hypothyroidic
- Active Rheumatoid Arthritis: Active Rheumatoid Arthritis meeting American College of Rheumatology (ACR) RA remission criteria
- Rheumatoid Arthritis in remission: Rheumatoid Arthritis in remission meeting American College of Rheumatology (ACR) RA remission criteria

SUMMARY:
RA is a chronic, autoimmune, inflammatory disease that involves small joints in the form of symmetrical polyarthritis and progresses with exacerbations and remissions. Pain, swelling, tenderness and morning stiffness are typical of the joints involved. Although it is approached as a primary joint disease, a wide variety of extra-articular involvements may also occur. In this cross sectional study sedimentation rate (ESR), C- Reactive protein (CRP), Tumor necrosis factor (TNF)-α, soluble-TNF-α receptor (TNF-R), Interleukin (IL)-1B and IL-10 were measured in three groups which were healthy volunteers, patients with RA in active period, and patients with RA in remission.

TNF-R can be the main pathophysiological factor and a marker showing activation. TNF-R can be very important in revealing the effect of TNF on the disease and the value of this effect in the treatment and ensuring the follow-up of the disease with CRP instead of ESR in activation.

DETAILED DESCRIPTION:
Aims: The etiopathogenesis of Rheumatoid Arthritis (RA) is not clearly understood. However, role of the cytokines takes an important part of this mechanism. The investigators aimed to bring a new approach to the concept of 'remission' in patients with RA.

Background: RA is a chronic, autoimmune, inflammatory disease that involves small joints in the form of symmetrical polyarthritis and progresses with exacerbations and remissions. Pain, swelling, tenderness and morning stiffness are typical of the joints involved. Although it is approached as a primary joint disease, a wide variety of extra-articular involvements may also occur. It is an interesting pathophysiological process, the exact cause of which is still unknown, with many environmental, genetic and potentially undiscovered possible factors in a chaotic manner.

Objective: In this prospective study, sedimentation rate (ESR), C- Reactive protein (CRP), Tumor necrosis factor (TNF)-α, soluble-TNF-α receptor (TNF-R), Interleukin (IL)-1B and IL-10 were measured in three groups which were healthy volunteers, patients with RA in active period, and patients with RA in remission. Disease activity score-28 (DAS-28) was calculated in active RA and RA in remission.

Methods: This study included 20 healthy volunteers, 20 remission patients with RA and 20 active RA patients. Venous blood samples were collected from patients in both healthy and RA groups.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals and Rheumatoid Arthritis patients meeting American College of Rheumatology (ACR) RA remission criteria.

Exclusion Criteria:

Smoking, Using Disease-Modifying Anti-Rheumatic Drugs (DMARD) and/or anti-inflammatory drugs other than cortisol and methotrexate, Receiving chemotherapy, Being hypothyroid

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included 20 healthy volunteers, 20 remission patients with RA and 20 active patients with RA. Patients who met the study criteria among patients with RA who applied to Maltepe University Medical Faculty Hospital Internal Medicine-Rheumatology Outpatient Clinic were included in the study
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
C Reactive Protein | up to 24 months
  Inflammatory biomarker
Erythrocyte sedimentation rate | up to 24 months
  Inflammatory biomarker
TNF alpha | up to 24 months
  Cytokine
DAS 28 | up to 24 months
  Disease activity scores
IL 1beta | up to 24 months
  Cytokine
IL 10 | up to 24 months
  Cytokine

CONTACTS AND LOCATIONS:
Overall Officials: Selim Nalbant, Prof, Principal Investigator — Maltepe University
Locations (1):
- Selim Nalbant, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malmstrom V, Catrina AI, Klareskog L. The immunopathogenesis of seropositive rheumatoid arthritis: from triggering to targeting. Nat Rev Immunol. 2017 Jan;17(1):60-75. doi: 10.1038/nri.2016.124. Epub 2016 Dec 5. PMID 27916980
- [Background] Deane KD, O'Donnell CI, Hueber W, Majka DS, Lazar AA, Derber LA, Gilliland WR, Edison JD, Norris JM, Robinson WH, Holers VM. The number of elevated cytokines and chemokines in preclinical seropositive rheumatoid arthritis predicts time to diagnosis in an age-dependent manner. Arthritis Rheum. 2010 Nov;62(11):3161-72. doi: 10.1002/art.27638. PMID 20597112
- [Background] Pratt AG, Isaacs JD. Seronegative rheumatoid arthritis: pathogenetic and therapeutic aspects. Best Pract Res Clin Rheumatol. 2014 Aug;28(4):651-9. doi: 10.1016/j.berh.2014.10.016. Epub 2014 Nov 18. PMID 25481556